CLINICAL TRIAL: NCT03948230
Title: Hypo-hydration, Mood and Cognition: the Effect of the Colour and Type of Drink
Brief Title: Hypo-hydration Mood and Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, David Benton, Professor, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DB-0519
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Mood; Cognitive Change
MeSH Terms: interventions — Salts

STUDY DESIGN:
Intervention Model Description: The study has six arms. Salt alone; salt plus water; salt plus colored water; placebo alone; placebo plus water; placebo plus colored water
Who Masked: Participant, Investigator
Masking Description: Salt / placebo will be consumed by capsule under a double-blind procedure
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sodium chloride / Water (Active Comparator): 300mg sodium chloride consumed in a capsule on two occasions with 300ml water
  Interventions: Biological: Salt with / without water
- Sodium chloride / no water (Active Comparator): 300 mg sodium chloride consumed
  Interventions: Biological: Salt with / without water
- Sodium chloride / colored water (Active Comparator): 300mg sodium chloride consumed in a capsule on two occasions with 300ml coloured water
  Interventions: Biological: Salt with / without water
- Placebo / water (Placebo Comparator): Placebo consumed in a capsule on two occasions with 300ml water
  Interventions: Biological: Salt with / without water
- Placebo / no water (Placebo Comparator): Placebo capsule consumed
  Interventions: Biological: Salt with / without water
- Placebo / coloured water (Placebo Comparator): Placebo consumed in a capsule on two occasions with 300ml colored water
  Interventions: Biological: Salt with / without water

INTERVENTIONS:
Biological: Salt with / without water — Drinks with and without a salt containing capsule

SUMMARY:
Recently changes in mood and cognition have been reported following minor reductions in hydration status. The aim is to explore that such changes in part at least reflect placebo response; therefore the consumption of plain or coloured water will be compared in drinks designed to differ in their ability to rehydrate.

DETAILED DESCRIPTION:
162 individuals will be subject to a temperature of 30°C for three hours, and mood and cognition monitored. Randomly on two occasions they will consume no drink or 300ml of plain or red colored water. In addition they will take a capsule containing sodium chloride or a placebo. Mood will be monitored using visual analogue scales and a battery of cognitive tests will be completed on three occasions: attention, episodic and working memory, reactions times. Urine osmolality will be measured at the beginning and end of the study and changes in body mass will be recorded. Changes in functioning will be related to the nature of the drink and changes in osmolality and body mass.

ELIGIBILITY:
Inclusion criteria:

* 18 to 30 years
* Non-smokers
* BMI < 30
* By self-report in good health
* Not taking medication for any psychological or other health disorder.

Exclusion Criteria:

* Do not meet inclusion criteria

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Mood rating: agreeable / hostile | Changes from baseline after 90 and 180 minutes
  A hundred millimetre lines will be anchored with the words agreeable/hostile and the subject will rate their mood by marking the line.. My measuring in millimetres a score between 0 and 100 will result with a higher score indicating a more positive mood.
Mood rating: confused / clearheaded | Changes from baseline after 90 and 180 minutes
  A hundred millimetre lines will be anchored with the words confused / clearheaded and the subject will rate their mood by marking the line.. My measuring in millimetres a score between 0 and 100 will result with a higher score indicating a more positive mood.
Mood rating: composed / anxious | Changes from baseline after 90 and 180 minutes
  A hundred millimetre lines will be anchored with the words composed / anxious and the subject will rate their mood by marking the line.. My measuring in millimetres a score between 0 and 100 will result with a higher score indicating a more positive mood.
Mood rating: depressed / elated | Changes from baseline after 90 and 180 minutes
  A hundred millimetre lines will be anchored with the words depressed / elated and the subject will rate their mood by marking the line.. My measuring in millimetres a score between 0 and 100 will result with a higher score indicating a more positive mood.
Mood rating: tired / energetic | Changes from baseline after 90 and 180 minutes
  A hundred millimetre lines will be anchored with the words tired / energetic and the subject will rate their mood by marking the line.. My measuring in millimetres a score between 0 and 100 will result with a higher score indicating a more positive mood.
Mood rating: confident / unsure | Changes from baseline after 90 and 180 minutes
  A hundred millimetre lines will be anchored with the words confident / unsure and the subject will rate their mood by marking the line.. My measuring in millimetres a score between 0 and 100 will result with a higher score indicating a more positive mood.

SECONDARY OUTCOMES:
Episodic memory | Changes from baseline after 90 and 180 minutes
  A list of 30 words will be presented after which the subject writes down as many as can be recalled. The resulting score will vary from 0-30.
Serial Sevens; test of working memory | Changes from baseline after 90 and 180 minutes
  28 numbers each of three digits will be presented and the subject indicates whether a subsequent number was exactly seven less. The measure reported is the response time in milli-seconds taken to respond
Attention: Arrow Flankers | Changes from baseline after 90 and 180 minutes
  A series is presented that can be >>>>> or >><>> and the subject has to indicated whether the middle symbol points to the right or left. The measure reported is the time taken to respond in milli-seconds
Reaction times | Changes from baseline after 90 and 180 minutes
  The time to press a button under an illuminated light was recorded in milli-seconds when there was 1, 2, 4, or 8 possible lamps that could be lit. 20 trials were performed with each of the four number of lights.

CONTACTS AND LOCATIONS:
Overall Officials: David Benton, DSc, Principal Investigator — Professor of Psychology
Locations (2):
- United Kingdom (2):
  - Psychology, Swansea University, Swansea, Wales
  - Swansea University, Swansea, Wales

IPD SHARING:
Plan to Share IPD: No